CLINICAL TRIAL: NCT01124487
Title: The Acute Effects of Oleic Acid Enriched-diets on Lipids, Insulin Sensitivity and Serum Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Dr. Kalanithi Nesaretnam, Malaysia Palm Oil Board
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: A001/09
Record Dates: First submitted 2010-05-12; First posted 2010-05-17 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Lipid Profile
Keywords: fat; inflammation; lipids; total cholesterol; Triglycerides; insulin sensitivity
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency; Inflammation; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- palm olein (Experimental)
  Interventions: Dietary Supplement: The acute effects of dietary fat on lipid profile, insulin sensitivity and inflammatory markers
- olive oil (Experimental)
  Interventions: Dietary Supplement: The acute effects of dietary fat on lipid profile, insulin sensitivity and inflammatory markers
- lard (Experimental)
  Interventions: Dietary Supplement: The acute effects of dietary fat on lipid profile, insulin sensitivity and inflammatory markers

INTERVENTIONS:
Dietary Supplement: The acute effects of dietary fat on lipid profile, insulin sensitivity and inflammatory markers

SUMMARY:
Objectives: To investigate the acute effects of olive oil, palm olein and lard on lipid profile, insulin sensitivity and inflammatory markers.

Hypothesis: Different dietary fats will alter lipid profile, insulin sensitivity and inflammatory markers postprandially.

DETAILED DESCRIPTION:
A randomized, single blind, crossover design was undertaken to test meals enriched with palm olein vs olive oil vs lard. Volunteers were asked to participate in three postprandial challenges, separated by at least 3-days. Subjects were provided a low fat meal(<10g fat) the day before the intervention. Fasting blood was collected the next day and the subjects were instructed to consume test meals (50g high fat meal). Further venous blood was collected at 30 min, 1h, 2h, 3h and 4h postprandially.

Primary outcome variable: Triacylglycerol (TAG) Secondary outcome variables: Insulin sensitivity (glucose, insulin), non esterified fatty acids (NEFA), inflammatory markers

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years
* BMI : 18.5-30 kg/m^2
* Healthy, men

Exclusion Criteria:

* medical history of cardiovascular disease, cancer, diabetes or chronic diseases
* BMI < 18.5 OR > 30 kg/m^2
* waist hip ratio > 0.9
* total cholesterol > 5.2 mmol/L
* triacylglycerol (TAG) > 2.2 mmol/L
* current use of antihypertensive or lipid lowering medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Triacylglycerol (TAG) | 4 h

SECONDARY OUTCOMES:
Insulin sensitivity (glucose, insulin), non-esterified fatty acids (NEFA), inflammatory markers | 4 h

CONTACTS AND LOCATIONS:
Overall Officials: Teng Kim Tiu, Msc, Principal Investigator — Malaysia Palm Oil Board and University of Malaya
Locations (1):
- Malaysian Palm Oil Board, Kajang, Selangor, Malaysia